CLINICAL TRIAL: NCT06416735
Title: Natriruetic Effect of Amiloride in Relation to the Alpha Adducin Gene (ADD-AMI) RS4961 Variant
Brief Title: Natriuretic Effect of Amiloride in Relation to the Alpha Adducin Gene (ADD-AMI) RS4961 Variant
Acronym: ADD-AMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Chiara Lanzani, medical doctor in nephrology unit, nephrologist, Ospedale San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ADD-AMI
Record Dates: First submitted 2023-09-04; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Hypertension Essential; Salt Excess; Genetic Hypertension
Keywords: Hypertension; Salt
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Amiloride

STUDY DESIGN:
Intervention Model Description: The study is a non-pharmacological interventional, single-center, national, non-randomised, comparative and open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- patients carrying the wild-type (GG) genotype of ADD1 rs4961 (Experimental): The protocol involves a test of oral administration of a single dose of Amiloride (5 or 10 mg based on body weight) to 20 patients carrying the wild-type (GG) genotype of ADD1 rs4961
  Interventions: Drug: Amiloride
- patients carriers of variant T (GT or TT) (Experimental): The test involves the administration of a single dose of 5 or 10 mg of Amiloride to 20 hypertensive carriers of the T variant (GT or TT)
  Interventions: Drug: Amiloride

INTERVENTIONS:
Drug: Amiloride — administration of a single dose of 5 or 10 mg of Amiloride (based on body weight) After oral intake of the drug, the increase in sodium in the urine ends within 8 hours

SUMMARY:
The study is a non-pharmacological interventional, single-center, national, non-randomised, comparative and open label.

DETAILED DESCRIPTION:
The study is carried out to evaluate primarily the difference in the activity of the renal transporter ENaC (through dosage of sodium) through its inhibition with a single dose of Amiloride in hypertensive patients characterized by the polymorphism of alpha Adducin rs496. It's also aimed to see the difference in potassium and the change in systolic and diastolic blood pressure after amiloride administration

ELIGIBILITY:
Inclusion Criteria:

* male patients aged 18-60 years;
* naïve hypertensive patients: newly diagnosed, never previously treated for hypertension;
* BMI<30 Kg/m2,
* documented first degree essential arterial hypertension (mean of the last 3 consecutive systolic BP measurements must be >=140 mmHg or diastolic BP >=90 mmHg;
* signature of the informed consent for participation in the study
* patient who has already undergone genomic DNA sampling (accompanied by relative consent) and genotyped for the ADD1 rs4961 variant (GG, GT or TT).

Exclusion Criteria:

known causes of secondary hypertension;

* severe or malignant hypertension; history of renal artery disease;
* significant renal disease (creatinine clearance less than 60 ml/min);
* hyperkalemia (Kpl > 6mEq/l) at enrollment visit;
* hypercalcaemia (Ca pl > 2.6 mmol/l) at enrollment visit;
* symptomatic hyperuricemia (> 7.5 mg/dl);
* liver disease (transaminases greater than 3 times the normal value);
* cardiac pathologies (myocardial infarction, atrial fibrillation, etc.);
* diabetes (fasting blood sugar >125mg/dl);
* in therapy with statins, NSAIDs, systemic steroids;
* known hypersensitivity to Amiloride or to any of the excipients;
* patients unable to express a valid consent -

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Evaluate urinary sodium | 3 hrs and 6 hrs
  Evaluation of sodium levels after oral administration of Amiloride

SECONDARY OUTCOMES:
Evaluate potassium levels | 3 hrs and 6 hrs
  Evaluation of potassium plasma levels after oral administration of Amiloride
Evaluation of systolic blood pressure | 3 hrs and 6 hrs
  Evaluation of systolic blood pressure after oral administration of Amiloride
Evaluation of diastolic blood pressure | 3 hrs and 6 hrs
  Evaluation of diastolic blood pressure after oral administration of Amiloride

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Lombardy, Italy